CLINICAL TRIAL: NCT01797939
Title: Predictive Factors of Response to Proton Pump Inhibitor Treatment in Patients With Gastroesophageal Reflux Disease Symptoms
Brief Title: Predictors of Proton Pump Inhibitor Response in Gastroesophageal Reflux Disease Patients
Status: Completed | Type: Observational
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Nayoung Kim, Professor, M.D., Seoul National University Bundang Hospital
Other Study IDs: B-1302-192-107
Record Dates: First submitted 2013-02-21; First posted 2013-02-25 (Estimated); Last update posted 2013-02-25 (Estimated); Status verified 2013-02

CONDITIONS: Erosive Reflux Disease; Non-erosive Reflux Disease; Functional Heartburn
Keywords: Erosive reflux disease (ERD); Non-erosive reflux disease (NERD); Functional heartburn (FH)
MeSH Terms: conditions — Non-Erosive Reflux Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Erosive reflux disease (ERD)
- Non-erovise reflux disease (NERD)
- Functional heartburn (FH)

SUMMARY:
Proton pump inhibitor (PPI) is widely used in patients with gastroesophageal reflux disease (GERD), however, some patients fail to respond to PPI therapy. Recent reporters suggest that depressive disorders, anxiety, sleep dysfunction were related with the symptomatic responses to a PPI treatments. Nevertheless, the predictive factors of response to PPI treatment still remain controversial. Therefore, the aims of this study were to investigate the efficacy of PPI therapy, and to evaluate the predictors of the PPI response in patients with symptomatic GERD by using the questionnaire which consisted of GERD symptoms, GERD impact scale (GIS), Epworth sleepiness scale (ESS), Pittsburgh sleep quality index (PSQI), Hospital anxiety and depression scale (HADS), and WHO quality of life scale abbreviated version (WHOQOL-BREF).

ELIGIBILITY:
Inclusion Criteria:

* Adult Subjects (From 16 to 85 years old)
* The participants with GERD symptoms were treated a PPI therapy.
* The participants completed a questionnaire. The questionnaire consisted of demographic data, GERD symptoms, GERD impact scale (GIS), Epworth sleepiness scale (ESS), Pittsburgh sleep quality index (PSQI), Hospital anxiety and depression scale (HADS), and WHO quality of life scale abbreviated version (WHOQOL-BREF).

Exclusion Criteria:

* Patients with a history of gastrointestinal surgery, Barrett's esophagus, esophageal motility disorder, peptic ulcer or gastroduodenal cancer and systemic disease requiring chronic medication (except for hypertension and diabetes mellitus) were excluded.
* Patients who took the PPI therapy less than 4 weeks were excluded.

Ages: 16 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Even the patients complain GERD symptoms such as heartburn and acid regurgitation the final diagnosis could be erosive reflux disease(ERD), non-erosive reflux disease (NERD) and even functional heartburn (FH).
Sampling Method: Non-Probability Sample
Enrollment: 197 (Actual)
Dates: Start 2008-07; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Efficacy of PPI therapy in these erosive reflux disease (ERD), non-erosive reflux disease (NERD), and functional heartburn (FH) groups | After 8 weeks of initial PPI administration
  Responses of dyspeptic symptoms were classified into 4 sections, as follows: complete response (more than 80% of symptom resolution), satisfactory response (symptoms remained less than 50%), partial response (symptoms remained for more than 50%), and refractory response (unresponsive to the eradication therapy). Then, the symptom responses were classified into 2 groups: responder with complete or satisfactory subgroup, and non-responder with partial or refractory responder subgroup.

SECONDARY OUTCOMES:
Predictors of the response to PPI treatment in patients with symptomatic GERD | After 8 weeks of initial PPI administration
  The participants were evaluated the predictors of PPI response by using the questionnaire which consisted of GERD symptoms, GERD impact scale (GIS), Epworth sleepiness scale (ESS), Pittsburgh sleep quality index (PSQI), Hospital anxiety and depression scale (HADS), and WHO quality of life scale abbreviated version (WHOQOL-BREF).

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea